CLINICAL TRIAL: NCT04083105
Title: Effectiveness of Nitrous Oxide Administration Prior to Intranasal Midazolam for Moderate Sedation in Pediatric Dental Patients
Brief Title: Nitrous Oxide Prior to Intranasal Midazolam for Moderate Dental Sedation in Pediatric Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospital Colorado (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Timothy Byrne, Regulatory Specialist, Children's Hospital Colorado
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-0404
Record Dates: First submitted 2019-08-16; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Dental Anxiety; Pain
Keywords: nitrous oxide; intranasal midazolam
MeSH Terms: conditions — Pain | interventions — Nitrous Oxide; Midazolam

STUDY DESIGN:
Intervention Model Description: Participants receiving moderate sedation for a dental procedure will be recruited and divided into one of two study arms.
Who Masked: Participant, Care Provider
Masking Description: Sedation provider who will administer the pain scale tests and the participant will be masked to the subject's assigned study arm (30% or 70% nitrous oxide with midazolam). The attending pediatric dentist and dental assistant will not be blinded for patient safety.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 30% Nitrous Oxide with Midazolam (Experimental): 30 percent nitrous oxide/70 percent oxygen will be administered for 5 minutes prior to intranasal midazolam.
  Interventions: Drug: Nitrous Oxide; Drug: Midazolam
- 70% Nitrous Oxide with Midazolam (Experimental): 70 percent nitrous oxide/30 percent oxygen will be administered for 5 minutes prior to intranasal midazolam.
  Interventions: Drug: Nitrous Oxide; Drug: Midazolam

INTERVENTIONS:
Drug: Nitrous Oxide — Nitrous oxide will be given prior to determine if it reduces pain from intranasal midazolam administration. Nitrous oxide is a minimal sedation drug used as an inhaled gas to reduce anxiety and produce anxiolysis and analgesia during dental procedures.
  Other Names: N2O
Drug: Midazolam — Intranasal midazolam will be given after nitrous oxide administration.
  Other Names: Versed

SUMMARY:
The purpose of this study is to assess the effectiveness of nitrous oxide/oxygen administration in reducing the discomfort of intranasal midazolam administration for moderate sedation for dental procedures.

DETAILED DESCRIPTION:
This study will determine the effectiveness of two different concentrations of nitrous oxide for reducing the pain of intranasal midazolam when given for subjects already planned for moderate sedation for completion of dental procedures in the pediatric dental clinic. Moderate dental sedation is useful because it helps relieve anxiety and make the dental procedure less memorable and more comfortable for the patient. Sedation appointments typically go smoothly when the patient is calm rather than when the patient is upset. Giving midazolam through the nose can be painful and the dental provider risks upsetting a patient and causing the sedation appointment to fail. Therefore, the goal of this study is to test whether nitrous oxide administration is effective in reducing the pain from intranasal midazolam administration. The effectiveness will be measured by the primary outcome of heart rate pre- and post- midazolam administration for the two randomly assigned study arms. The first study arm will be given 30% nitrous/70% oxygen and the second study arm will be given 70% nitrous/30% oxygen prior to the midazolam administration. The secondary outcome will compare subject, dental provider, and the parent/guardian answers to questions regarding the subject's experience pre- and post- midazolam administration. The investigators hypothesize lower changes in heart rate and less pain reported following midazolam administration in subjects given 70% nitrous oxide.

ELIGIBILITY:
Inclusion Criteria:

* Patients selected to undergo moderate sedation at the Children's Hospital Colorado Dental Clinic
* Subject must have visited the dental clinic within 4 months of their sedation appointment for a regular dental examination
* Subject must have a well-child visit with their primary care physician within the last 12 months prior to their sedation appointment
* Child must fall between the ages of 3 to 8 years old
* Child must be healthy, American Society of Anesthesiologists scale I or II
* Children under 4 years will be asked to count and explain the instrument before enrollment.

Exclusion Criteria:

* Upper respiratory illness (URI) symptoms less than 4 weeks before sedation appointment
* American Society of Anesthesiologists scale III or IV
* Children with special needs including intellectual disability, congenital malformations, chronic conditions
* Chronic lung disease
* Cyanotic heart disease
* Children with anatomic airway abnormalities or moderate to severe tonsillar hypertrophy
* Any contraindications to nitrous oxide use including: Chronic obstructive pulmonary diseases, current upper respiratory tract infections, recent middle ear disturbance/surgery, severe emotional disturbances or drug-related dependencies, previous treatment with bleomycin sulfate, methylenetetrahydrofolate reductase (MTHFR) deficiency, cobalamin (Vitamin B12) deficiency
* Allergy or hypersensitivity to nitrous oxide or midazolam

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2019-07-12 (Actual); Primary Completion 2021-07-11 (Estimated); Study Completion 2021-07-11 (Estimated)

PRIMARY OUTCOMES:
Heart rate | through the study completion, an average of 2 years
  Measured in beats per minute with range from 50-190 bpm. A great change in heart rate indicates more pain and less effect of the nitrous oxide. Heart rate is an autonomic reflex to determine the effect of mental and physical stressors including painful stimuli. The participants resting heart rate will be compared to the heart rate immediately after intranasal midazolam administration for a change in heart rate value.

SECONDARY OUTCOMES:
Visual analog scales (VAS) for pain | through the study completion, an average of 2 years
  Scale from 1 (no pain) to 10 (most possible pain). A higher score indicates greater pain. VAS will be obtained from the subjective standpoint of the parent/guardian of the parent and the dental provider during time points before and after the administration of intranasal midazolam.
Visual analog scales (VAS) for fear | through the study completion, an average of 2 years
  Scale from 1 (no fear) to 10 (very fearful). A higher score indicates greater fear. VAS will be obtained from the subjective standpoint of the parent/guardian of the parent and the dental provider during time points before and after the administration of intranasal midazolam.
Wong-Baker Faces scale for pain | through the study completion, an average of 2 years
  Scale from 0 (no hurt) to 10 (hurts worst). A higher score indicates more pain. Wong-Baker Faces scale will be recorded from the subjective standpoint of the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Chin, DDS, MS, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual personal data with other researchers.